CLINICAL TRIAL: NCT05910359
Title: Ultrasound Prediction of Persistent Occiput Posterior Position in Active Labor: a Multicentric Prospective Cross-sectional Study
Brief Title: Ultrasound Prediction of POPP in Active Labor
Acronym: (POPP-UP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Familiari Alessandra, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5830
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Labor Complication; Fetal Head to Enter Pelvic Brim; Failure, Affecting Fetus or Newborn
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Multicenter prospective cross-sectional interventional study without drug nor device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persistent Occiput Posterior Position (Experimental): transabdominal and transperineal ultrasound by expert sonographers
  Interventions: Diagnostic Test: Ultrasound
- Anterior Occiput Position at delivery (Active Comparator): transabdominal and transperineal ultrasound by expert sonographers
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — transabdominal and transperineal ultrasound by expert sonographers

SUMMARY:
Persistent occiput posterior position (POPP) represents a relevant risk factor for various adverse outcomes: prolonged labor, higher incidence of operative delivery and/or cesarean section for non-reassuring fetal conditions, higher incidence of high-grade perineal tears (OASIS). For such reasons, labor with POPP needs particular and non-routinary attention.

Hence, it is important to diagnose in advance fetuses who present POPP to assure more adequate assistance in labor. Furthermore, digital examination shows a lower detection rate for such condition if compared to ultrasound in labor.

This multicenter prospective cross-sectional interventional study aims to evaluate the occiput position and the descent of the fetal head at the beginning of active labor to predict POPP at delivery. All the participants will be subjected to transabdominal and transperineal ultrasound at the beginning of active labor (between 3 and 8 cm of cervical dilatation) to evaluate the position of the fetal head and its descent. At the delivery, the position of the fetal head and the features of the second stage of the labor will be recorded.

DETAILED DESCRIPTION:
Background and rationale Occiput posterior position (OP) is the most common fetal malposition during labor. Such anomaly shows a correlation with higher risk of operative delivery and cesarean section, prolonged labor duration, neonatal morbidity, high-grade perineal lacerations. It is estimated that around 15-30% of fetuses in cephalic presentation start the labor in OP. Of these, 10-15% remain OP at full cervical dilatation, but only 5-8% remains in persistent OP position (POPP) at delivery, especially in nulliparous women.

The importance of knowing the precise position of the fetal head is related to the possible adverse outcome that POPP carries, requiring adequate surveillance during labor and delivery. The non-routinary surveillance consist of:

* Continuous non intermittent monitoring of fetal wellbeing (with cardiotocography)
* Rationalization of peridural anesthesia doses, due to prolonged labor
* Maternal position during labor facilitating descent and rotation of the fetal head
* Active cure of the perineum to reduce the risk of high-grade perineal tears.

In case of operative delivery, knowing the exact position of the fetal occiput ensure a better positioning of the vacuum extractor.

Ultrasound in labor ward demonstrated a higher performance compared to routine care (vaginal examination) in diagnosing fetal occiput position. Various approaches have been described to induce fetal head rotation: manual or instrumental intrauterine attempts, or maternal position changes (without any strong evidence).

The mechanism of POPP remains unclear. Predisposing factors are several: nulliparity, android pelvis, obesity, fetal macrosomia, preterm birth7. Some authors suggest that the presence of fibroids, uterine adherences or analgesia in labor could affect the overall risk of malpositions. Relatively to anesthesia, some authors suggest that the prolonged second stage of labor could be the reason for a higher incidence of POPP in women undergoing peridural procedures. Studies evaluating the rotation of the fetal head during labor progression reported discordant results. Some authors suppose that POPP is secondary to an OP at the beginning of the labor, others that anterior or transverse position can be modified by already mentioned risk factors.

In a study conducted on a population of 918 women in labor reported how the main part of OP fetuses at the beginning of labor will rotate to OA at birth, while cases of POPP are related to a persistence of posterior position rather than a malrotation. Eggebo et al reported that the main part of women presenting POPP at birth showed different occiput position at the time of rupture of membranes, reinforcing the theory of malrotation. Another multicentric study, on a population of 100 women, reported no cases of POPP in fetuses with OA at the beginning of labor. Furthermore, evaluating the spine position, the authors say that in case of OP and posterior spine, one case out of seven rotates in OA at birth.

Studies about prediction of POPP show heterogeneity, small populations and in some cases exclusion of participants in case of cesarean section or operative deliveries. Moreover, the grade of descent of the fetal head is a fundamental information not always considered, unlike cervical dilatation, for diagnosis of active labor.

OBJECTIVES

Primary Objective Primary objective of the study is to evaluate POPP in the study population.

Secondary Objectives To develop a predictive model for diagnose POPP at the beginning of active labor.

METHODS Study design Multicenter prospective cross-sectional interventional study without drug nor device Population We will enroll all pregnant women with diagnosis of active labor, admitted to delivery room, afferent to the to the participating centers, satisfying the following inclusion criteria.

Study duration The study will last 12 months. Inclusion criteria

* Age ≥18 y.o.;
* Pregnant women with diagnosis of active labor, admitted to delivery room;
* Singleton;
* At term (>37 weeks);
* Cephalic presentation;
* Signed written informed consent to study participation. Exclusion criteria
* Age <18 y.o.;
* Preterm deliveries;
* Multiple pregnancies;
* Elective cesarean section;
* Non-cephalic presentation;
* Incomplete obstetrical data;
* Refusal to provide informed consent.

Variables and procedures For each participant, several anamnestic data will be recorded at the enrollment. Each participant, after written consent, once in active labor (defined as cervical dilatation between 4 and 8 cm with presence of regular and painful uterine contractions) will undergo transabdominal and transperineal ultrasound by expert sonographers. Data about fetal occiput position, fetal eyes visualization and fetal head descent (measured by Angle of Progression) will be recorded. Then, at the delivery, we will evaluate the position of the fetal head at birth and the features of the second stage of the labor. All neonatal clinical characteristics will be collected.

At the enrollment, after consent, the following data will be recorded:

* Demographic and anthropometric data (i.e., age (y), ethnicity, height (m), weight (kg), BMI);
* Parity
* Gestational Age (weeks + days)
* Cervical dilatation (cm)
* Type of labor (spontaneous, induced)
* Membrane integrity

Then, all the participants will undergo a transabdominal and transperineal US in lithotomic position to evaluate:

* Fetal occiput position (anterior, transverse, posterior) (Fig.1)
* In case of posterior occiput, women will be divided in two groups according to the number of visible eyes (one-eye vs two-eyes, Fig. 2)
* Fetal spine position (anterior, transverse, posterior)
* Angle of progression (AoP) described as the angle between the long axis of the pubic bone and a line from the lowest edge of the pubis drawn tangential to the deepest bony part of the fetal skull.

After the birth, following data will be collected:

* Type of birth (spontaneous, operative vaginal, cesarean sections CS)
* Position at birth
* Eventual anesthesia
* Kristeller manouver
* Episiotomy or perineal tears
* Active phase duration (min) and Second stage duration (min);
* Sex and weight of the baby;
* APGAR score at 1 and 5 minutes
* Cord blood samples (pH and Base Excess, arteriosus and venous)
* Eventual NICU admission.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18 y.o.;

  * Pregnant women with diagnosis of active labor, admitted to delivery room;
  * Singleton;
  * At term (>37 weeks);
  * Cephalic presentation;
  * Signed written informed consent to study participation.

Exclusion Criteria:

* • Age <18 y.o.;

  * Preterm deliveries;
  * Multiple pregnancies;
  * Elective cesarean section;
  * Non-cephalic presentation;
  * Incomplete obstetrical data;
  * Refusal to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 593 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
the incidence of POPP in the study population | 1 year
  How many POPP in labor

IPD SHARING:
Plan to Share IPD: No